CLINICAL TRIAL: NCT01701700
Title: The Effectiveness of Portable Electronic Vision Enhancement Systems (EVES) in Comparison to Optical Magnifiers for Near Vision Activities in Visual Impairment - The p-EVES Study
Brief Title: The Effectiveness of Portable Electronic Vision Enhancement Systems (p-EVES) for Near Vision in Visual Impairment
Acronym: p-EVES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Manchester University NHS Foundation Trust (Other Government)
Collaborators: National Institute for Health Research, United Kingdom (Other Government); University of Manchester (Other); Cardiff University (Other); Bangor University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PB-PG-0211-24105; R01715 (Other: CMFT)
Record Dates: First submitted 2012-10-01; First posted 2012-10-05 (Estimated); Last update posted 2018-12-04 (Actual); Status verified 2018-11

CONDITIONS: Moderate or Severe Vision Impairment, Both Eyes
Keywords: portable electronic magnifiers
MeSH Terms: conditions — Lymphoma, Follicular; Vision Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- portable electronic magnifier (Experimental): Use of a prescribed electronic magnifier plus existing optical aids for a period of 2 months
  Interventions: Procedure: portable electronic magnifier; Procedure: optical aids
- optical aids (Active Comparator): Use of existing optical aids for 2 months
  Interventions: Procedure: optical aids

INTERVENTIONS:
Procedure: portable electronic magnifier
  Other Names: electronic video magnifier; portable CCTV; electronic vision enhancement system; EVES
  Arms: portable electronic magnifier
Procedure: optical aids
  Other Names: magnifiers

SUMMARY:
Over 1 million people in the UK suffer from untreatable visual impairment, many of them elderly. The major complaint of visually impaired people is their inability to carry out simple tasks, especially those involving reading. It is known that this activity limitation is a major cause of depression in an older population, and it is reflected in reduced quality of life. Low vision clinics, mostly based within hospital ophthalmology departments, dispense optical magnifiers to allow patients to carry out these tasks again, but these devices do have limitations (unusual posture, short working distance, monocular viewing). Although electronic magnifiers have been around since the 1960s, they were initially very large and expensive. Recent advances in technology have brought about an explosion in the number and range of portable and moderately-priced aids, which can be used binocularly, in a natural working position: these are currently not available through the NHS. Evidence is needed as to whether these portable hand-held electronic magnifiers could offer a significant benefit to the majority of patients, and therefore whether they should be routinely dispensed in low vision clinics.

The proposed study is a two-arm randomised crossover trial with existing users of optical magnifiers being assigned to use a hand-held electronic magnifier in addition to their existing devices for 2 months. Reading and task performance will be measured with the aid, and compared to the performance with optical aids, and the patient will be asked to report on the comparisons between the aids.

ELIGIBILITY:
Inclusion Criteria:

* Patients of Manchester Royal Eye Hospital
* Visual impairment secondary to range of stable ocular pathologies (no change in VA > 2 lines in previous 6 months)
* Currently possess a near vision optical magnifying device.
* VA <= 6/30 (<=0.7 logMAR) and/or log contrast sensitivity <=1.20

Exclusion Criteria:

* Current use of personal EVES device
* Hearing inadequate to respond to verbal instruction
* Habitual language not English
* A physical disability preventing the participant from operating the device
* A score of less than 19 on the Mini-Mental State Examination

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2013-02; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
usage of magnifiers | Change from baseline at 2 months and 4 months
  Use of Manchester Low Vision Questionnaire to quantify device usage
reading speed | Change from baseline at 2 months and 4 months
  Reading speed using the device assessed by MNREAD test

SECONDARY OUTCOMES:
speed of performance of activities of daily living | Change from baseline at 2 months and 4 months
  total time taken to performance 5 selected activities of daily living using aids if required
difficulty with near vision activities | Change from baseline at 2 months and 4 months
  Use of NV-VFQ-15 questionnaire to self-rate difficulty in performance of near vision activities
health related quality of life | Change from baseline at 2 months and 4 months
  Use of EQ-5D and VISQOL questionnaires to self-rate health-related quality of life
well-being | Change from baseline at 2 months and 4 months
  use of WHO-5 questionnaire to self-rate wellbeing

CONTACTS AND LOCATIONS:
Overall Officials: Chris M Dickinson, PhD, Principal Investigator — University of Manchester
Locations (1):
- Manchester Royal Eye Hospital, Manchester, United Kingdom